CLINICAL TRIAL: NCT03624712
Title: Prospective, Tricentric Open Trial on the Analysis and Optimization of Predictive and Therapeutic Models in Uterine Neoplasms
Brief Title: Analysis and Optimization of Predictive and Therapeutic Models in Uterine Neoplasms
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University Hospital Heidelberg (Other); University of Homburg (Other); University Hospital Freiburg (Other)
Responsible Party: Sponsor
Other Study IDs: ZGynO_DENOVA
Record Dates: First submitted 2018-07-04; First posted 2018-08-10 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Uterine Neoplasms
MeSH Terms: conditions — Uterine Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- uterine neoplasms: Women with operable and inoperable uterine malignomas (cervical cancer, endometrial cancer, uterine sarcoma)
  Interventions: Diagnostic Test: uterine neoplasms

INTERVENTIONS:
Diagnostic Test: uterine neoplasms — Analysis of circulating (CTC) and disseminating tumor cells (DTC), determination of Human Papilloma Virus (HPV), Douglas cytology, DNA analysis in blood, proteome analysis, sentinel lymph node detection

SUMMARY:
Evaluation of clinical, therapeutic and prognostic relevance of new experimental results as well as optimization of therapeutic models and development of a new algorithm for therapeutic plan and therapy in patients with uterine neoplasm

ELIGIBILITY:
Inclusion Criteria:

* Confirmed uterine malignancy ( cervical cancer, endometrial cancer, sarcoma)
* If operable: surgical primary therapy: laparoscopic/robot-assisted or open radical gyneco-oncological surgery
* Written consent
* Willingness and ability to participate in all study-specific procedures
* Age ≥ 18 years

Exclusion Criteria:

* Severe and acute general disease in the last 4 weeks
* Acute or chronic psychiatric disorders
* Other factors questioning study participation (e.g. acute psychosocial stress, insufficient understanding of nature and consequences of the study, inadequate skills of the German language)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with operable or inoperable uterine malignancy (cervical cancer, endometrial cancer, sarcoma)
Sampling Method: Non-Probability Sample
Enrollment: 580 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
CTC and DTC analysis | 12 months
  Counting the number of tumor cells in blood and bone marrow
HPV | 12 months
  Analysis of HPV types by DNA tests in peripheral blood, bone marrow, sentinel-lymph node, cervical-, endometrial- and myometrial-tissue, intraperitoneal wash fluid
DNA | 12 months
  Determination of DNA in peripheral blood
Douglas cytology | 12 months
  Intraperitoneal wash fluid
Proteomic analysis | 12 months
  Analysis of proteins by mass spectrometry in removed uterine and sentinel lymph node tissue
Sentinel lymph nodes | 12 months
  Number of detectable lymph nodes by Tc99m- and indocyanine green-labeling
Peripheral nerve conduction velocity | 12 months
  Intra- and interindividual comparison of N. obturatorius, N. pudendus between pre an post radical gynecological surgery
Urodynamic- cystomanometry between pre an post radical gynecological surgeryuroflowmetry | 12 months
  pressur/volume relationship
CTC and DTC analysis | 12 months
  Identification and quantification of genetic variants and mutations
Urodynamic- urethral pressure profile between pre an post radical gynecological surgeryuroflowmetry | 12 months
  cm H20
Urodynamic- uroflowmetry between pre an post radical gynecological surgeryuroflowmetry | 12 months
  rate of flow of urine

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tuebingen, Department of Women's Health, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No